CLINICAL TRIAL: NCT00317733
Title: A Double-Blind, Placebo-Controlled Evaluation of Safety and Efficacy of Epicutaneously Applied IDEA-033 (Ketoprofen in Transfersome) in Comparison to Oral Celecoxib for the Treatment of Pain Associated With Osteoarthritis of the Knee
Brief Title: Ketoprofen in Transfersome Compared to Oral Celecoxib and Placebo for Pain Associated With Osteoarthritis of the Knee
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: IDEA AG (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CL-033-II-03; NCT01309464 (obsolete NCT alias)
Record Dates: First submitted 2006-04-21; First posted 2006-04-25 (Estimated); Last update posted 2009-03-20 (Estimated); Status verified 2009-03

CONDITIONS: Osteoarthritis, Knee
Keywords: Ketoprofen; Transfersome; Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Ketoprofen

INTERVENTIONS:
Drug: Ketoprofen in Transfersome

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of 110 mg ketoprofen in Transfersome applied to the skin twice daily as compared to placebo and oral celecoxib 200 mg per day for the relief of signs and symptoms of osteoarthritis of the knee for a period of six weeks.

DETAILED DESCRIPTION:
This is a multicenter, randomized (patients are assigned different treatments based on chance), double-blind (neither the patient nor the physician knows whether drug or placebo is being taken, or at what dosage), double-dummy, parallel group, placebo- and active-controlled study to determine the safety and effectiveness of 110 mg of ketoprofen in Transfersome, applied to the skin, in subjects experiencing at least moderate pain when not taking analgesic medication secondary to osteoarthritis pain of the knee. The study hypothesis is that ketoprofen in Transfersome applied to the skin twice daily will be more effective than placebo for the relief of the signs and symptoms of osteoarthritis of the knee as measured by the Visual Analog Scale (VAS) of the Western Ontario and McMaster Universities Index (WOMAC) pain, WOMAC function and subject global asessment of response to therapy at Week 6. WOMAC is a questionaire consisting of 24 questions designed to assess the three dimensions of pain, disability and joint stiffness in osteoarthritis of the knee. Safety evaluations include reports of adverse events, laboratory tests and skin irritation.

Patients will receive one of the following treatments for six weeks - 110 mg ketoprofen in Transfersome applied to the skin twice per day plus one placebo capsule administered orally twice per day, 100 mg celecoxib administered orally twice per day plus placebo Transfersome applied to the skin twice per day, Placebo Transfersome applied to the skin twice per day plus one placebo capsule administered orally twice twice per day.

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthritis of the knee for a minimum of six months
* Patient´s rating of pain in the index knee while not taking oral NSAIDs of at least 3 using a 5-point Likert scale
* Presenting two out of the three following criteria - Morning stiffness of less than 30 minutes duration, Crepitus on motion, Age >= 40 years
* Patients must have used oral NSAIDs at least 3 days per week for the 3 months prior to screening or the patient was taking an NSAID on a regular basis (>25 out of 30 days) at a therapeutic level for at least 30 days prior to screening
* Each of the following three criteria (the osteoarthritis flare criteria) must be met - Index knee pain assessment at walking at least 40 mm on VAS at baseline, Increase of index knee pain at walking by at least 15 mm on VAS at baseline compared to screening, Physician´s global assessment of osteoarthritis 3-5 and at least 1 grade increase from screening

Exclusion Criteria:

* Grade 1 or Grade 4 severity of the index knee based on Kellgren and Lawrence radiographic criteria
* Intraarticular injections or arthroscopy of the index knee within 3 months prior to screening
* Signs of any clinically important inflammation of the index knee including redness, warmth and or a large bulging effusion with the loss of normal contour
* Crystalline-induced synovitis in the index knee
* History, physical examination or radiographic suggestive of acute inflammatory arthritis, rheumatoid arthritis, psoriatic arthritis, septic arthritis, gout, pseudogout, fibromyalgia, lupus erythematosus, or other types of inflammatory arthritis of the index knee

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360
Dates: Study Completion 2004-01

PRIMARY OUTCOMES:
Change from baseline at Week 6 on the VAS version of the WOMAC pain subscale; Change from baseline at Week 6 on the VAS version of the WOMAC function subscale; Subject global assessment of response to therapy measured on a 5-point Likert scale at Week 6

SECONDARY OUTCOMES:
Change from baseline at Weeks 2 and 4 for WOMAC pain and physical function scores; Subject global assessment of response to therapy at Weeks 2 and 4; Physician's global assesment of osteoarthritis at Weeks 2, 4 and 6

CONTACTS AND LOCATIONS:
Overall Officials: McNeil Consumer & Specialty Pharmaceuticals Clinical Trial, Study Director — McNeil Consumer & Specialty Pharmaceuticals, a Division of McNeil-PPC, Inc.

REFERENCES:
- [Result] Rother M, Lavins BJ, Kneer W, Lehnhardt K, Seidel EJ, Mazgareanu S. Efficacy and safety of epicutaneous ketoprofen in Transfersome (IDEA-033) versus oral celecoxib and placebo in osteoarthritis of the knee: multicentre randomised controlled trial. Ann Rheum Dis. 2007 Sep;66(9):1178-83. doi: 10.1136/ard.2006.065128. Epub 2007 Mar 15. PMID 17363401